CLINICAL TRIAL: NCT00833248
Title: A Randomised, Parallel Arm, Open-label Trial Comparing Degarelix With Goserelin Plus Anti-androgen Flare Protection (Bicalutamide), in Terms of Prostate Size Reduction in Prostate Cancer Patients of Intermediate-to-high Risk, Who Require Neoadjuvant Hormone Therapy Prior to Radiotherapy (Curative Intent)
Brief Title: Neoadjuvant Study Investigating Degarelix in Patients Suffering From Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS30; 2008-005232-33 (EudraCT Number)
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Results first posted 2012-09-27 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Degarelix 240 mg/80 mg (Experimental): The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The second and third doses of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections on Days 28 and 56, respectively.
  Interventions: Drug: Degarelix
- Goserelin (3.6 mg) + bicalutamide (50 mg) (Active Comparator): On Day 0, the participants began once-daily oral (p.o.) treatment with bicalutamide as anti-androgen flare protection. This treatment continued for 2 weeks after the first dose of goserelin (i.e. 17 days in total).
  On Day 3, the first goserelin implant was inserted s.c. into the abdominal wall. The second and third doses of goserelin were administered on Days 31 and 59, respectively.
  Interventions: Drug: Goserelin; Drug: Bicalutamide

INTERVENTIONS:
Drug: Degarelix — The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The second and third doses of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections on Days 28 and 56, respectively.
  Other Names: FE200486; Firmagon
  Arms: Degarelix 240 mg/80 mg
Drug: Goserelin — Goserelin implants (3.6 mg) were inserted s.c. into the abdominal wall every 28 days. The first dose was administered on Day 3. The second and third doses of goserelin were administered on Days 31 and 59, respectively.
  Other Names: Zoladex
  Arms: Goserelin (3.6 mg) + bicalutamide (50 mg)
Drug: Bicalutamide — On Day 0, participants began once-daily per-oral (p.o.) treatment with bicalutamide (50 mg) as anti-androgen flare protection; this treatment continued for 14 days after the first dose of goserelin.
  Other Names: Casodex
  Arms: Goserelin (3.6 mg) + bicalutamide (50 mg)

SUMMARY:
The purpose of this phase 3B trial was to see how well a new trial drug (degarelix) works in terms of reducing the size of the prostate volume in prostate cancer patients who were scheduled to undergo subsequent radiotherapy for treatment of their prostate cancer. Prior to receiving radiotherapy, it is recommended that patients with intermediate to high risk prostate cancer are pre-treated with hormone therapy (so-called neoadjuvant therapy) which is known to reduce the size of the prostate and thereby decrease the required radiation field and enable a more safe and effective treatment. In this trial, participants were randomly selected (like flipping a coin) to receive either degarelix given alone or a standard hormone therapy (combination of goserelin and bicalutamide. The treatment was given for three months and the prostate size was measured by ultra sound at the beginning and at the end of the trial. The participants were required to come to the clinic for 5 or 6 visits during the three months.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent before any trial-related activity is performed.
* Has a confirmed prostate cancer in which this type of treatment is needed.

Exclusion Criteria:

* Previous treatment for prostate cancer
* Previous trans-urethral resection of the prostate
* Patients who are lymph node positive or have other metastatic disease
* Use of urethral catheter
* Current treatment with a 5-alpha reductase inhibitor or α-adrenoceptor antagonist.
* History of severe untreated asthma, anaphylactic reactions, or severe urticaria and/or angioedema.
* Hypersensitivity towards any component of the investigational product
* Other previous cancers within the last five years with the exception of prostate cancer and some types of skin cancer.
* Certain risk factors for abnormal heart rhythms/QT prolongation (corrected QT interval over 450 msec., Torsades de Pointes or use of certain medications with potential risk)
* Clinical disorders other than prostate cancer including but not limited to renal, haematological, gastrointestinal, endocrine, cardiac, neurological, psychiatric disease, alcohol or drug abuse or other conditionals as judged by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (66):
- United States (19):
  - Alabama Research Center, Birmingham, Alabama
  - Urology Centers of Alabama, Homewood, Alabama
  - Alaska Urological Association, Anchorage, Alaska
  - Arizona Urologic Specialists, Tuscon, Arizona
  - Orange County Urology, Lagua Hills, California
  - Tri-Valley Urology Medical Group, Murrieta, California
  - Connecticut Clinical Research Center, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - DCT -Celebration, LLC dba Discovery Clinical Trials, Celebration, Florida
  - Pinellas Urology Inc., St. Petersburg, Florida
  - Palm Beach Urology Associates, Wellington, Florida
  - Summit Research Institute, Bloomington, Indiana
  - Northeast Indiana Research, Fort Wayne, Indiana
  - Urology Center Research Institute, Englewood, New Jersey
  - Urology Group of New Mexico, Albuquerque, New Mexico
  - Premier Medical Group of Hudson, Baldwinsville, New York
  - University Urology Associates, New York, New York
  - Urology Associates, Nashville, Tennessee
  - Urology of Virginia, Norfolk, Virginia
- France (19):
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - CHU Henri Mondor, Créteil
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital de la Timone, Marseille
  - CRLC Val d'Aurelle Oncology Radiotherapy, Montpellier
  - Hôpital Tenon, Paris
  - Hôpital Saint Louis, Radiotherapy Departement, Paris
  - Clinique Francheville, Périgueux
  - CHU La Milétrie, Oncology Radiotherapy, Poitiers
  - Clinique Saint Brieuc, Saint-Brieuc
  - Centre de Lutte Contre le Cancer Nantes-Atlantique Centre René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Centre de radiologie Saint Louis, Toulon
  - Clinique du Parc, Toulouse
  - IGR, Villejuif
- Germany (4):
  - Charité-Universitätsmedizin, Campus Benjamin Franklin Klinik für Urologie, Berlin
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Universitätsklinikum Dresden, Klinik und Poliklinik für Urologie, Dresden
  - Universitätsklinikum Ulm, Klinik für Strahlentherapie und Radioonkologie, Ulm
- Greece (4):
  - General University Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens, "Sismanogleio", University of Athens, Marouse, Athens
  - University General Hospital of Loannina, Medical School, Loannina
  - University General Hospital of Patras, Pátrai
- Netherlands (6):
  - Albert Schweitzer Ziekenhuis, Ioc., Dordwijk, Dordrecht
  - Groene Hart Ziekenhuis, urology, Gouda
  - Franciscus Gasthuis, Dept. urology, Rotterdam
  - Maastad Ziekenhuis, Ioc. Clara, Rotterdam
  - Vlietland Ziekenhuis, Dept. urology, Schiedam
  - St. Elisabeth Ziekenhuis Tilburg, Tilburg
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Fundación IVO, Valencia
- United Kingdom (10):
  - Kent Oncology Centre Maidstone Hospital, Maidstone, Kent
  - Mount Vernon Cancer Center, Northwood, Middlesex
  - Oncology Royal United Hospital Bath NHS Trust, Bath
  - Addenbrooke's Hospital, Oncology Centre, Cambridge
  - St. James' University Hospital, Leeds
  - The Royal Marsden NHS, Foundation Trust, London
  - Charing Cross Hospital, London
  - Northern Centre for Cancer Treatment, Newcastle General Hospital, Newcastle upon Tyne
  - Southhampton General Hospital, Cancer Care Directorate, Southhampton Oncology Centre, Southhampton
  - Velindre Hospital, Cardiff University, Whitchurch

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976
- [Derived] Mason M, Maldonado Pijoan X, Steidle C, Guerif S, Wiegel T, van der Meulen E, Bergqvist PB, Khoo V. Neoadjuvant androgen deprivation therapy for prostate volume reduction, lower urinary tract symptom relief and quality of life improvement in men with intermediate- to high-risk prostate cancer: a randomised non-inferiority trial of degarelix versus goserelin plus bicalutamide. Clin Oncol (R Coll Radiol). 2013 Mar;25(3):190-6. doi: 10.1016/j.clon.2012.09.010. Epub 2012 Dec 17. PMID 23257248

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited by outpatient urologists, radiotherapists or oncologists. A total of 240 patients were to be randomised in a 3:1 ratio to one of two treatment groups (180 participants were to be treated with degarelix; 60 participants were to be treated with goserelin+bicalutamide). The recruitment period was April 2009 - June 2011.
Period: Overall Study
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Started | 181 | 65
Full Analysis Set (FAS) | 180 | 64
Per Protocol (PP) Analysis Set | 164 | 57
Safety Analysis Set | 181 | 64
Completed | 177 | 62
Not Completed | 4 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg) | Total
Number analyzed (Participants) | 180 | 64 | 244
Age Continuous [Mean (Standard Deviation); unit: years] — Full analysis set (FAS).
  years | 70.6 (6.37) | 70.8 (5.96) | 70.6 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants] — FAS.
  Participants
    Female | 0 | 0 | 0
    Male | 180 | 64 | 244
Race (NIH/OMB) [Count of Participants; unit: Participants] — FAS.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 15 | 3 | 18
    White | 163 | 61 | 224
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — FAS.
  participants
    United States | 45 | 16 | 61
    France | 60 | 22 | 82
    Greece | 5 | 2 | 7
    Spain | 9 | 3 | 12
    Netherlands | 11 | 2 | 13
    Germany | 9 | 4 | 13
    United Kingdom | 41 | 15 | 56
Body Weight [Mean (Standard Deviation); unit: kilogram] — FAS.
  kilogram | 83.6 (14.2) | 80.9 (12.4) | 82.9 (13.8)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] — FAS.
  kilogram per square meter | 27.8 (3.99) | 26.8 (3.69) | 27.5 (3.93)
Gleason Score [Number; unit: participants] — FAS. The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    Gleason Score 2-6 | 41 | 12 | 53
    Gleason Score 7 | 97 | 42 | 139
    Gleason Score 8-10 | 42 | 10 | 52
Stage of Prostate Cancer [Number; unit: participants] — FAS. Prostate cancer stage was classified according to the Tumor, Nodes, and Metastatic (TNM) scale to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor. Some participants did not have their prostate cancer classified for the complete TNM scale (9 participants).
  participants
    Localized | 111 | 41 | 152
    Locally Advanced | 63 | 20 | 83
    Metastatic | 0 | 0 | 0
    Not Classifiable | 6 | 3 | 9
Serum Testosterone Levels [Median (Full Range); unit: nanograms per milliliter] — FAS.
  nanograms per milliliter | 3.92 [0.557 to 11.2] | 4.42 [0.188 to 8.16] | 4.06 [0.188 to 11.2]
Serum Prostate-Specific Antigen (PSA) Levels [Median (Full Range); unit: nanograms per millilter] — FAS.
  nanograms per millilter | 10 [2.5 to 339] | 9.75 [2.9 to 80] | 9.95 [2.5 to 339]
Serum Oestradiol Levels [Median (Full Range); unit: nanograms per deciliter] — FAS.
  nanograms per deciliter | 1.9 [0.74 to 4.4] | 1.9 [1 to 3.6] | 1.9 [0.74 to 4.4]
Prostate Volume [Mean (Standard Deviation); unit: milliliter] — FAS. Prostate volume was measured with a Trans Rectal Ultrasound Scan (TRUS).
  milliliter | 50.9 (20.3) | 52.5 (18.8) | 51.3 (19.9)
Total International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: scores on a scale] — FAS. The IPSS is a tool commonly used to assess the severity of lower urinary tract symptoms (LUTS), and to monitor the progress of the disease once treatment has been initiated. The participant completes a questionnaire containing 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Each question is assigned a score of 0-5. The total score is then classified according to the following scale: 0 to 7 = mildly symptomatic; 8 to 19 = moderately symptomatic; and 20 to 35 = severely symptomatic.
  scores on a scale | 9.5 (6.71) | 8.46 (6.3) | 9.23 (6.61)
Quality of Life (QoL) Related to Urinary Symptoms [Mean (Standard Deviation); unit: scores on a scale] — FAS. The IPSS questionnaire included an additional single question to assess the participant's QoL in relation to his urinary symptoms. The question was: 'If you were to spend the rest of your life with your urinary condition the way it is now, how would you feel about that?' The possible answers to this question ranged from 'delighted' (a score of '0') to 'terrible' (a score of '6').
  scores on a scale | 2.27 (1.63) | 1.94 (1.56) | 2.19 (1.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Prostate Size Based on Trans Rectal Ultra Sound (TRUS) at Week 12 (Full Analysis Set)
Description: TRUS is a method of measuring the size of the prostate.
Time Frame: After treatment of 12 weeks compared to Baseline
Population: FAS, Observed Case (OC) i.e. only participants with a reported value were included in the analysis.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 176 | 62
milliliter | -36.0 (14.5) | -35.3 (16.7)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); FAS. Estimates from analysis of variance with treatment as factors and baseline IPSS and baseline Prostate volume as covariates; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be established if the treatment difference in adjusted (for baseline volume, and baseline total IPSS) mean percentage reduction was significantly greater (two-sided at α=0.05 level) than Δ = 10 points (non-inferiority margin) in both the FAS and PP analyses sets; p = 0.8942, ANCOVA; The baseline IPSS and baseline Prostate volume were used as covariates and treatment was used as a factor in the analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-4.74 to 4.14]

2. Primary Outcome: Change From Baseline in Prostate Size Based on Trans Rectal Ultra Sound (TRUS) at Week 12 (Per Protocol Analysis Set)
Description: TRUS is a method of measuring the size of the prostate.
Time Frame: After treatment of 12 weeks compared to Baseline
Population: FAS, OC.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 154 | 54
milliliter | -36.2 (14.5) | -35.4 (16.9)
Statistical Analysis 1: Comparison: Degarelix 240 mg/80 mg vs Goserelin (3.6 mg) + Bicalutamide (50 mg); PP analysis set. Estimates from analysis of variance with treatment as factors and baseline IPSS and baseline Prostate volume as covariates; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9123, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.268, 95% CI 2-sided [-5.05 to 4.52]

3. Secondary Outcome: Change From Baseline in Total International Prostate Symptom Score (IPSS) at Week 4, 8, and 12
Description: The IPSS is a tool commonly used to assess the severity of lower urinary tract symptoms (LUTS), and to monitor the progress of the disease once treatment has been initiated. The participant completes a questionnaire containing 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Each question is assigned a score of 0-5. The total score is then classified according to the following scale: 0 to 7 = mildly symptomatic; 8 to 19 = moderately symptomatic; and 20 to 35 = severely symptomatic.
Time Frame: After treatment of 4, 8, and 12 weeks compared to Baseline
Population: FAS, OC.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 177 | 63
scores on a scale
  Week 4 | -0.21 (5.05) | 0.36 (4.83)
  Week 8 | -1.53 (5.43) | 0.02 (5.41)
  Week 12 | -1.71 (5.54) | 0.11 (5.13)

4. Secondary Outcome: Change From Baseline in Serum Testosterone Levels During the Study
Time Frame: After treatment of 4, 8, and 12 weeks compared to Baseline
Population: FAS, OC.
Measure: Median (Full Range); unit: nanograms per milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 170 | 63
nanograms per milliliter
  Week 4 | -3.8 [-11.06 to -0.51] | -4.22 [-8.06 to 0.52]
  Week 8 | -3.77 [-11.01 to -0.51] | -4.26 [-8.11 to -0.14]
  Week 12 | -3.81 [-11.09 to -0.51] | -4.3 [-8.11 to -0.14]

5. Secondary Outcome: Change From Baseline in Serum Prostate-Specific Antigen (PSA) Levels During the Study
Time Frame: After treatment of 4, 8, and 12 weeks compared to Baseline
Population: FAS, OC.
Measure: Median (Full Range); unit: nanograms per milliliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 172 | 62
nanograms per milliliter
  Week 4 | -6.3 [-333 to 4.5] | -5.9 [-76 to 4]
  Week 8 | -7.95 [-337 to -2] | -8.8 [-79.4 to -1.7]
  Week 12 | -8.35 [-338 to -2] | -9.05 [-78.8 to -1.8]

6. Secondary Outcome: Change From Baseline in Serum Oestradiol Levels During the Study
Time Frame: After treatment of 4, 8, and 12 weeks compared to Baseline
Population: FAS, OC.
Measure: Median (Full Range); unit: nanogram per deciliter
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 124 | 36
nanogram per deciliter
  Week 4 | -1.55 [-4.35 to -0.63] | -1.65 [-3.5 to -0.9]
  Week 8 | -1.6 [-3.6 to -0.27] | -1.65 [-3.55 to -0.95]
  Week 12 | -1.55 [-4.35 to -0.48] | -1.6 [-3.55 to -0.8]

7. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Related to Urinary Symptoms at Each Visit
Description: The IPSS questionnaire included an additional single question to assess the participant's QoL in relation to his urinary symptoms. The question was: 'If you were to spend the rest of your life with your urinary condition the way it is now, how would you feel about that?' The possible answers to this question ranged from 'delighted' (a score of '0') to 'terrible' (a score of '6').
Time Frame: After treatment of 4, 8, and 12 weeks compared to Baseline
Population: FAS, OC.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 179 | 63
scores on a scale
  Week 4 | -0.07 (1.31) | 0.16 (0.92)
  Week 8 | -0.24 (1.34) | 0.05 (1.11)
  Week 12 | -0.33 (1.46) | 0.16 (1.4)

8. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The table presents the number of participants with normal baseline and at least one post-baseline markedly abnormal value.
Time Frame: Baseline to 12 weeks of treatment
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 181 | 64
participants
  Diastolic blood pressure <=50 and decrease >=15 | 0 | 0
  Diastolic blood pressure >=105 and increase >=15 | 3 | 0
  Systolic blood pressure <=90 and decrease >=20 | 0 | 0
  Systolic blood pressure >=180 and increase >=20 | 1 | 1
  Heart rate <=50 and decrease >=15 | 1 | 1
  Heart rate >=120 and increase >=15 | 0 | 0
  Body weight decrease of >=7 percent | 3 | 2
  Body weight increase of >=7 percent | 5 | 0

9. Secondary Outcome: Number of Participants With Markedly Abnormal Values in Safety Laboratory Variables
Description: The figures present the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) levels of safety laboratory variables. Only the laboratory variables that had at least one percentage of participants in either group with abnormal value are presented, more variables were included in the study.
Time Frame: Baseline to 12 weeks of treatment
Population: Safety analysis set.
Measure: Number; unit: participants
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Number analyzed (Participants) | 181 | 64
participants
  B-Haematocrit (Ratio) <=0.37 | 31 | 8
  B-Haemoglobin (g/L) <=115 | 4 | 1
  S-Alanine aminotransferase (IU/L) >3 x ULN | 1 | 1
  S-Potassium (mmol/L) >=5.8 | 4 | 1
  S-Urea nitrogen (mmol/L) >=10.7 | 10 | 3

ADVERSE EVENTS:
Time Frame: 12 weeks.
Description: Each participant's condition was monitored throughout the trial from the time of signing the informed consent until the end of the follow-up period. The investigator was to record all adverse events (AEs) in the AE log of the participant's Case Report Form.
Arm/Group | Degarelix 240 mg/80 mg | Goserelin (3.6 mg) + Bicalutamide (50 mg)
Serious Adverse Events (participants affected / at risk) | 7/181 | 0/64
Other Adverse Events (participants affected / at risk) | 158/181 | 53/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/80 mg (N=181) | Goserelin (3.6 mg) + Bicalutamide (50 mg) (N=64)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/80 mg (N=181) | Goserelin (3.6 mg) + Bicalutamide (50 mg) (N=64)
Injection site pain (General disorders) | 60 (93) | 1 (1)
Injection site erythema (General disorders) | 45 (73) | 0 (0)
Asthenia (General disorders) | 13 (15) | 6 (6)
Injection site pruritus (General disorders) | 13 (19) | 0 (0)
Fatigue (General disorders) | 11 (13) | 6 (6)
Injection site swelling (General disorders) | 11 (17) | 0 (0)
Libido decreased (Psychiatric disorders) | 12 (12) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 11 (13) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 14 (15) | 7 (7)
Hot flush (Vascular disorders) | 108 (132) | 40 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.